CLINICAL TRIAL: NCT03238482
Title: Pharmacokinetic Study Comparing Salmeterol/Fluticasone Easyhaler 50/250 µg/Dose Products and Seretide Diskus 50/250 µg/Dose in Healthy Subjects
Brief Title: Comparing Salmeterol/Fluticasone Easyhaler and Seretide Diskus (SAIMI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3106012
Record Dates: First submitted 2017-07-11; First posted 2017-08-03 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Seretide Diskus (Active Comparator): salmeterol-fluticasone 2 inhalations as a single dose
  Interventions: Drug: salmeterol-fluticasone
- Salmeterol/fluticasone Easyhaler, E (Experimental): salmeterol-fluticasone 2 inhalations as a single dose
  Interventions: Drug: salmeterol-fluticasone
- Salmeterol/fluticasone Easyhaler, F (Experimental): salmeterol-fluticasone 2 inhalations as a single dose
  Interventions: Drug: salmeterol-fluticasone
- Salmeterol/fluticasone Easyhaler, G (Experimental): salmeterol-fluticasone 2 inhalations as a single dose
  Interventions: Drug: salmeterol-fluticasone

INTERVENTIONS:
Drug: salmeterol-fluticasone — Seretide Diskus 50/250 µg/dose
  Arms: Seretide Diskus
Drug: salmeterol-fluticasone — Salmeterol/fluticasone Easyhaler 50/250 µg/dose, product E
  Arms: Salmeterol/fluticasone Easyhaler, E
Drug: salmeterol-fluticasone — Salmeterol/fluticasone Easyhaler 50/250 µg/dose, product F
  Arms: Salmeterol/fluticasone Easyhaler, F
Drug: salmeterol-fluticasone — Salmeterol/fluticasone Easyhaler 50/250 µg/dose, product G
  Arms: Salmeterol/fluticasone Easyhaler, G

SUMMARY:
The purpose of this study is to compare absorption of salmeterol and fluticasone from Salmeterol/fluticasone Easyhaler test products to the commercially available product Seretide Diskus

ELIGIBILITY:
Main inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Males and females, 18-60 (inclusive) years of age.
3. Normal weight defined as body mass index (BMI) 19-30 kg/m2 (BMI = weight/height2).
4. Weight at least 50 kg.

Main exclusion Criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic, endocrine, neurological or psychiatric disease.
2. Any condition requiring regular concomitant treatment.
3. Any clinically significant abnormal laboratory value or physical finding that in the opinion of the investigator may interfere with the interpretation of study results or constitute a health risk for the subject if he/she takes part in the study.
4. Known hypersensitivity to the active substance(s) or the lactose.
5. Pregnant or lactating females and females of childbearing potential not using proper contraception.
6. Blood donation or loss of significant amount of blood within 90 days prior to first study treatment administration.
7. Administration of another investigational medicinal product within 90 days prior to first study treatment administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of salmeterol | between 0-34 hours after dosing
  Cmax of salmeterol
Peak plasma concentration (Cmax) of fluticasone propionate | between 0-34 hours after dosing
  Cmax of fluticasone propionate
Area under the plasma concentration versus time curve (AUC) of salmeterol | 0-34 hours after dosing
  AUC from time zero to the last sample with the quantifiable concentration
Area under the plasma concentration versus time curve (AUC) of fluticasone propionate | 0-34 hours after dosing
  AUC from time zero to the last sample with the quantifiable concentration
Truncated area under the plasma concentration versus time curve (AUC) of salmeterol | 0-30 minutes after dosing
  AUC from time zero to 30 min after study treatment administration

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of salmeterol | 0-34 hours after dosing and extrapolation
  AUC from time zero to infinity
Area under the plasma concentration versus time curve (AUC) of fluticasone propionate | 0-34 hours after dosing and extrapolation
  AUC from time zero to infinity
The time to reach the maximum concentration (tmax) of salmeterol | 0-34 hours after dosing
  tmax of salmeterol
The time to reach the maximum concentration (tmax) of fluticasone propionate | 0-34 hours after dosing
  tmax of fluticasone propionate
The terminal elimination half-life (t1/2) of salmeterol | 0-34 hours after dosing
  t1/2 of salmeterol
The terminal elimination half-life (t1/2) of fluticasone propionate | 0-34 hours after dosing
  t1/2 of fluticasone propionate

OTHER OUTCOMES:
Adverse events | through study completion, an average of 6 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Sairanen, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Clinical Pharmacology Unit, Orion Pharma, Espoo, Finland